CLINICAL TRIAL: NCT01879358
Title: Randomized Comparison of a Sirolimus Eluting ORSIRO Stent With a Biolimus-eluting NOBORI Stent in Patients Treated With Percutaneous Coronary Intervention
Brief Title: Sirolimus Eluting ORSIRO Stent Versus Biolimus-eluting NOBORI Stent
Acronym: SORT OUT VII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Lisette Okkels Jensen, MD DMSci PhD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SORT OUT VII; OUH (Other: Odense University Hospital)
Record Dates: First submitted 2013-03-18; First posted 2013-06-17 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
Keywords: Drug-eluting stent; Safety; Efficacy
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ORSIRO stent (Active Comparator): ORSIRO stent group
  Interventions: Device: Drug-eluting stent
- NOBORI stent (Active Comparator): NOBORI stent group
  Interventions: Device: Drug-eluting stent

INTERVENTIONS:
Device: Drug-eluting stent
  Other Names: ORSIRO sirolimus-eluting stent; NOBORI biolimus-eluting stent

SUMMARY:
The aim of the Danish Organization for Randomized Trials with Clinical Outcome (SORT OUT) is to compare the safety and efficacy of the sirolimus eluting ORSIRO stent and the biolimus-eluting NOBORI stent in a population-based setting, using registry detection of clinically driven events

DETAILED DESCRIPTION:
SORT OUT VII is a randomized, multicenter, all-comer, two-arm, non-inferiority trial comparing the sirolimus eluting ORSIRO stent to the biolimus-eluting NOBORI stent in treating atherosclerotic coronary artery lesions.

Primary Endpoint:

Target lesion failure within 12 months of stent implantation (combination of cardiac death, myocardial infarction (not index procedure related) not related to other than index lesion or target lesion revascularization).

Secondary Endpoints:

Individual components of the primary end point comprised the secondary end points and stent thrombosis rate according to the Academic Research Consortium definition (see protocol for further specification of secondary endpoints).

Clinically driven event detection will be used to avoid study-induced reinterventions. Data on mortality, hospital admission, coronary angiography, repeat percutaneous coronary intervention, and coronary bypass surgery will be obtained for all randomly allocated patients from the following national Danish administrative and healthcare registries: the Civil Registration System; the Western Denmark Heart Registry; the Danish National Registry of Patients, which maintains records on all hospitalizations in Denmark; and the Danish Registry of Causes of Death

Inclusion criteria:

at least 18 years old chronic stable coronary artery disease or acute coronary syndromes at least one coronary artery lesion with more than 50% diameter stenosis requiring treatment with a drug-eluting stent

Exclusion criteria:

life expectancy of less than one year allergy to aspirin, clopidogrel, sirolimus, or biolimus participation in another randomized trial nability to provide written informed consent

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or over with chronic stable coronary artery disease or acute coronary syndromes, and at least one coronary artery lesion with more than 50% diameter stenosis, requiring treatment with a drug-eluting stent. There are no restrictions on number of treated lesions, number of treated vessels, or lesion length.

Exclusion Criteria:

* Exclusion criteria are life expectancy of less than one year; an allergy to aspirin, clopidogrel, ticagrelor, prasugral, sirolimus, or biolimus; participation in another randomized trial; or inability to provide written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2314 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-02 (Actual); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac death, myocardial infarction or target lesion revascularization | 12 months
  Target lesion failure within 12 months of stent implantation (combination of cardiac death, myocardial infarction (not index procedure related) not related to other than index lesion or target lesion revascularization)

SECONDARY OUTCOMES:
Cardiac death, myocardial infarction, target lesion revascularization, target vessel revascularization, all cause mortality, stent thrombosis | 12 months
  Cardiac mortality Myocardial infarction Target lesion revascularization Target vessel revascularization All cause mortality Stent thrombosis rate according to the Academic Research Consortium definition Secondary endpoints will be assessed after 1 year, 2 years, 3 years, 4 years and 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jens F Lassen, MD DMSci, Study Chair — Aarhus University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Jensen LO, Thayssen P, Hansen HS, Christiansen EH, Tilsted HH, Krusell LR, Villadsen AB, Junker A, Hansen KN, Kaltoft A, Maeng M, Pedersen KE, Kristensen SD, Botker HE, Ravkilde J, Sanchez R, Aaroe J, Madsen M, Sorensen HT, Thuesen L, Lassen JF; Scandinavian Organization for Randomized Trials With Clinical Outcome IV (SORT OUT IV) Investigators. Randomized comparison of everolimus-eluting and sirolimus-eluting stents in patients treated with percutaneous coronary intervention: the Scandinavian Organization for Randomized Trials with Clinical Outcome IV (SORT OUT IV). Circulation. 2012 Mar 13;125(10):1246-55. doi: 10.1161/CIRCULATIONAHA.111.063644. Epub 2012 Feb 3. PMID 22308301
- [Derived] Troan J, Christiansen EH, Hansen KN, Eftekhari A, Jakobsen L, Maeng M, Freeman P, Jensen RV, Christensen MK, Noori M, Ellert-Gregersen J, Stottrup NB, Kahlert J, Veien KT, Jensen LO. Five-year outcomes of patients with diabetes mellitus treated with a sirolimus-eluting or a biolimus-eluting stents with biodegradable polymer. From the SORT OUT VII trial. Diab Vasc Dis Res. 2024 Sep-Oct;21(5):14791641241283939. doi: 10.1177/14791641241283939. PMID 39311502
- [Derived] Hansen KN, Jensen LO, Maeng M, Christensen MK, Noori M, Kahlert J, Jakobsen L, Junker A, Freeman P, Ellert-Gregersen J, Raungaard B, Terkelsen CJ, Veien KT, Christiansen EH. Five-Year Clinical Outcome of the Biodegradable Polymer Ultrathin Strut Sirolimus-Eluting Stent Compared to the Biodegradable Polymer Biolimus-Eluting Stent in Patients Treated With Percutaneous Coronary Intervention: From the SORT OUT VII Trial. Circ Cardiovasc Interv. 2023 Jan;16(1):e012332. doi: 10.1161/CIRCINTERVENTIONS.122.012332. Epub 2023 Jan 17. PMID 36649389
- [Derived] Jensen LO, Thayssen P, Maeng M, Ravkilde J, Krusell LR, Raungaard B, Junker A, Terkelsen CJ, Veien KT, Villadsen AB, Kaltoft A, Tilsted HH, Hansen KN, Aaroe J, Kristensen SD, Hansen HS, Jensen SE, Madsen M, Botker HE, Berencsi K, Lassen JF, Christiansen EH. Randomized Comparison of a Biodegradable Polymer Ultrathin Strut Sirolimus-Eluting Stent With a Biodegradable Polymer Biolimus-Eluting Stent in Patients Treated With Percutaneous Coronary Intervention: The SORT OUT VII Trial. Circ Cardiovasc Interv. 2016 Jul;9(7):e003610. doi: 10.1161/CIRCINTERVENTIONS.115.003610. PMID 27412869
- [Derived] Jensen LO, Thayssen P, Maeng M, Ravkilde J, Hansen HS, Jensen SE, Botker HE, Berencsi K, Lassen JF, Christiansen EH. Randomized comparison of a sirolimus-eluting Orsiro stent with a biolimus-eluting Nobori stent in patients treated with percutaneous coronary intervention: Rationale and study design of the Scandinavian Organization for Randomized Trials with Clinical Outcome VII trial. Am Heart J. 2015 Aug;170(2):210-5. doi: 10.1016/j.ahj.2015.05.009. Epub 2015 May 22. PMID 26299216
- See also: SORT OUT IV with same clinically event driven methodology — http://www.ncbi.nlm.nih.gov/pubmed/22308301